CLINICAL TRIAL: NCT05018169
Title: Behavioral Activation for Treatment of Depression in Adolescents With Autism Spectrum Disorder: A Pilot Study
Brief Title: Behavioral Activation for Treatment of Depression in Adolescents With Autism
Acronym: BA-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Micah Mazurek, Novartis U.S. Foundation Professor of Education, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR200385
Record Dates: First submitted 2021-08-03; First posted 2021-08-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Depression; Autism
MeSH Terms: conditions — Depression; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BA-A (Experimental): Teens will participate in BA-A. BA-A is a 12-session manualized treatment that utilizes established BA strategies and incorporates common mental health treatment adaptations for young people with ASD.
  Interventions: Behavioral: BA-A

INTERVENTIONS:
Behavioral: BA-A — Session 1 focuses on the treatment rationale, structure, and expectations, and includes psychoeducation on depression. Session 2 focuses on working with parent(s) to help them support their teen through treatment. Session 3 focuses on the (situation)/behavior/feeling cycle and how teens individuals can get trapped in a cycle of depression and inactivity. Session 4 focuses on the assessment of values and choosing preferred activities to target. Session 5 focuses on teaching skills for in-person and electronic communication. Session 6 focuses on identifying barriers to treatment success. Session 7 focuses on teaching teens to handle disagreements. Session 8 focuses on the utilization of adaptive coping skills. Sessions 9-11 are meant to be used flexibly and should include review of any challenging concepts. Session 12 is the termination session and focuses on maintaining treatment gains. Between every session, teens will track their activity for homework.

SUMMARY:
In this study, the investigators will examine the feasibility, acceptability, and preliminary efficacy of a novel, behavior-based approach for treatment of depression symptoms in adolescents with autism spectrum disorder or ASD (i.e., Behavioral Activation for Adolescents with ASD, BA-A).

DETAILED DESCRIPTION:
In this study, the investigators will examine the feasibility, acceptability, and preliminary efficacy of a novel, behavior-based approach for treatment of depression symptoms in adolescents with ASD (i.e., Behavioral Activation for Adolescents with ASD, BA-A). BA-A is a 12-session manualized treatment that utilizes established behavioral activation strategies and incorporates common mental health treatment adaptations for young people with ASD. For this project, the investigators will pilot BA-A with 23 adolescents (12-17 years of age) with ASD and clinically significant depression symptoms. To investigate BA-A feasibility, the investigators will examine treatment session attendance and therapist treatment fidelity. To investigate BA-A acceptability, the investigators will utilize a mixed methods approach, inclusive of surveys and qualitative interviews, to inform BA-A protocol refinement. To investigate BA-A preliminary efficacy, the investigators will examine depression symptoms, as well as secondary outcome measures, at pre-treatment, post-treatment, and one-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of ASD by a qualified health care provider
* Children's Depression Inventory, Second Edition (CDI2) parent-report and/or self-report T- score ≥ 65
* Wechsler Abbreviated Scale of Intelligence, Second Edition (WASI-II) Full Scale IQ, Two-Subtest Form (FSIQ-2) ≥ 85
* Participation of a parent or legal guardian living in the same home who can read and write in English at or above the fifth grade level
* Teens must have been on a stable dose of medications for mood, anxiety, or behavior for at least three months prior to enrollment and have no planned medication changes during study period
* Not actively participating in another psychotherapy during study period

Exclusion Criteria:

* High suicide risk
* Physical aggression
* Psychotic and/or manic symptoms

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Children's Depression Inventory, Second Edition, Parent Report | Change from pre-treatment to post-treatment (i.e., within one week of finishing 12-week treatment) and one-month following treatment
Children's Depression Inventory, Second Edition, Self Report | Change from pre-treatment to post-treatment (i.e., within one week of finishing 12-week treatment) and one-month following treatment
Children's Depression Rating Scale, Revised | Change from pre-treatment to post-treatment (i.e., within one week of finishing 12-week treatment) and one-month following treatment

SECONDARY OUTCOMES:
Spence Children's Anxiety Scale, Self Report | Change from pre-treatment to post-treatment (i.e., within one week of finishing 12-week treatment) and one-month following treatment
Spence Children's Anxiety Scale, Parent Report | Change from pre-treatment to post-treatment (i.e., within one week of finishing 12-week treatment) and one-month following treatment
Social Skills Improvement System, Parent Report | Change from pre-treatment to post-treatment (i.e., within one week of finishing 12-week treatment) and one-month following treatment

OTHER OUTCOMES:
Treatment Fidelity Checklists | Within 3 months of treatment completion
  Treatment Fidelity Checklists will be completed by trained research assistants not involved in the implementation of the intervention.
Acceptability/Satisfaction Surveys and Interviews, Self Report | Post-treatment (i.e., within one week of finishing 12-week treatment)
Acceptability/Satisfaction Surveys and Interviews, Parent Report | Post-treatment (i.e., within one week of finishing 12-week treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No